CLINICAL TRIAL: NCT01136915
Title: A Phase IV Pilot Study to Evaluate Kidney Damage Measured by Neutrophil Gelatinase-Associated Lipocalin (NGAL) as a New Bio-Marker in Patients With Severe Fall in eGFR Undergoing Percutaneous Coronary Intervention With IOPAMIDOL Injection 370 or IODIXANOL 320
Brief Title: Kidney Damage In Patients With Severe Fall In eGFR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IOP-118
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Stenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Iopamidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IOPAMIDOL injection 370 (Active Comparator)
  Interventions: Drug: Iopamidol 370
- Iodixanol 320 (Active Comparator)
  Interventions: Drug: Iodixanol 320

INTERVENTIONS:
Drug: Iopamidol 370 — one time administration for PCI
  Other Names: Isovue 370
  Arms: IOPAMIDOL injection 370
Drug: Iodixanol 320 — Iodixanol 320 single injection for percutaneous coronary injection
  Arms: Iodixanol 320

SUMMARY:
This is a pilot study using a randomized, double blinded, comparison of two iodinated contrast agents used during percutaneous coronary intervention (PCI). All patients enrolled must have and estimated glomerular filtration [eGFR] < 30 mL/min/1.73 m2. Statistical summaries will be presented to analyse the various laboratory tests for the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Provides written Informed Consent
* Is at least 18 years of age;
* Is scheduled for or likely to undergo percutaneous coronary intervention;
* Has documented estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m2 calculated with the MDRD formula within 72 hours prior the enrolment.

Exclusion Criteria:

* Is a pregnant or lactating female
* Has a history of severe congestive heart failure
* Has a history of hyperthyroidism
* Has unstable renal function
* Has a history of hypersensitivity to iodinated contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institu De Cardiologie De Montreal, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Iopamidol 370: Iopamidol 370: Non-ionic low-osmolar iodinated contrast media: single administration for percutaneous coronary intervention procedure
- Iodixanol 320: Iodixanol 320 Non-ionic iso-osmolar iodinated contrast media comparator: single administration for percutaneous coronary intervention procedure
Period: Overall Study
Arm/Group | Iopamidol 370 | Iodixanol 320
Started | 8 | 7
Completed | 6 | 6
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Exclusion criterion met | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Iopamidol 370: Iopamidol 370: Non-ionic low-osmolar iodinated contrast media: single intravenous administration for percutaneous coronary intervention procedure; dose was limited to the minimum volume required to achieve diagnostic information and/or guide therapeutic intervention.
- Iodixanol 320: Iodixanol 320 Non-ionic iso-osmolar iodinated contrast media comparator: single intravenous administration for percutaneous coronary intervention procedure; dose was limited to the minimum volume required to achieve diagnostic information and/or guide therapeutic intervention.
- Total: Total of all reporting groups
Arm/Group | Iopamidol 370 | Iodixanol 320 | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (9.1) | 67.7 (14.2) | 68.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 1 | 4
  China | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Impact on the Trajectory of Serum and Urinary NGAL Following the Administration of Non-ionic, Low-osmolar Contrast Media in Comparison to a Non-ionic, Iso-osmolar Contrast Media.
Description: Mean change from baseline values for serum NGAL at 2,4,6,24,48, and 72 hours, and urine NGAL at 2,4,6,24, and 48 hours following the administration of contrast media.
Time Frame: Baseline and 2,4,6,24, 48, and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Iopamidol 370 Serum NGAL: Serum NGAL (ng/mL) mean change from baseline at 2,4,6,24,48, and 72 hours post-administration of iopamidol 370
- Iopamidol 370 Urine NGAL: Urine NGAL (ng/mL) mean change from baseline at 2,4,6,24,and 48 hours post-administration of iopamidol 370
- Iodixanol 320 Serum NGAL: Serum NGAL (ng/mL) mean change from baseline at 2,4,6,24,48, and 72 hours post-administration of iodixanol 320
- Iodixanol 320 Urine NGAL: Urine NGAL (ng/mL) mean change from baseline at 2,4,6,24,and 48 hours post-administration of iodixanol 320
Arm/Group | Iopamidol 370 Serum NGAL | Iopamidol 370 Urine NGAL | Iodixanol 320 Serum NGAL | Iodixanol 320 Urine NGAL
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL
  2 hours post-dose | -33.03 (26.24) | -12.24 (54.13) | -103.23 (45.63) | -29.51 (55.67)
  4 hours post-dose | -6.39 (33.26) | -29.98 (50.98) | -102.53 (65.80) | -52.09 (65.31)
  6 hours post-dose | 13.03 (32.60) | -10.81 (26.01) | -45.53 (101.85) | -51.00 (65.46)
  24 hours post-dose | 38.76 (79.94) | 22.51 (61.31) | -20.13 (76.28) | -20.75 (36.89)
  48 hours post-dose | 28.08 (83.99) | 37.78 (35.34) | -90.34 (79.20) | 30.09 (106.75)
  72 hours post-dose | -16.88 (33.76) | NA (NA) — Urine NGAL not measured at 72 hours post-dose as per protocol. | -25.89 (161.56) | NA (NA) — Urine NGAL not measured at 72 hours post-dose as per protocol.

ADVERSE EVENTS:
Arm/Group | Iopamidol 370 | Iodixanol 320
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days